CLINICAL TRIAL: NCT02794948
Title: Chinese Medicine(Hu Yang Yang Kun Formula) for Primary Ovarian Insufficiency:Randomized, Double-blind, DHEA-controlled Trial
Brief Title: Chinese Medicine(Hu Yang Yang Kun Formula) for Primary Ovarian Insufficiency
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Guangzhou University of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: YN2014TS06
Record Dates: First submitted 2016-03-19; First posted 2016-06-09 (Estimated); Last update posted 2018-04-10 (Actual); Status verified 2016-03

CONDITIONS: Primary Ovarian Insufficiency
Keywords: primary ovarian insufficiency; TCM intervention
MeSH Terms: conditions — Primary Ovarian Insufficiency | interventions — Dehydroepiandrosterone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Chinese Medicine intervention (Experimental): Chinese medicine HuYang Yang Kun Formula 1 capsule every time per day for 3 day per month, DHEA(dehydroepiandrosterone) placebo 1 sack every time, twice a day for three months
  Interventions: Other: Chinese medicine granules (HuYang Yang Kun Formula)
- Western intervention (Active Comparator): DHEA(dehydroepiandrosterone) 1 sack every time twice a day for three months. Chinese medicine formula granules placebo 1 capsule every time per day for 3 day per month.
  Interventions: Dietary Supplement: dehydroepiandrosterone

INTERVENTIONS:
Other: Chinese medicine granules (HuYang Yang Kun Formula) — Take Chinese medicine granules (HuYang Yang Kun Formula), 1 sack every time,twice a day Take DHEA(dehydroepiandrosterone) placebo,1 capsule every time ,once a day. Treatment for 3 months Both Chinese Medicine formula granules and DHEA placebo were produced by Jiangyin Medical &pharmaceutical limited company in Jiangsu province
  Arms: Chinese Medicine intervention
Dietary Supplement: dehydroepiandrosterone — The DHEA( dehydroepiandrosterone)25mg,1 capsule every time once a day. Take Chinese medicine granules placebo , 1 sack every time,twice a day Treatment is 3 months. DHEA were produced by General Nutrition Center(GNC)company in America and The placebo granules of Chinese Medicine were produced by Jiangyin Medical &pharmaceutical limited company in Jiangsu province.
  Arms: Western intervention

SUMMARY:
The purpose of this research is providing valuable traditional chinese medicine theory and formula in treating Primary Ovarian insufficiency.

DETAILED DESCRIPTION:
Primary ovarian insufficiency is a problem that is to be solved urgently in the field of reproductive endocrine. According to the basic theory of traditional Chinese Medicine and clinical experience, investigators developed a Chinese medicine formula(Hu yang yang kun,Hyyk). This research is designed according to the principle of randomized double blind control and evaluated the effectiveness and safety of Hyyk, hope to provide a kind of effective medicine in treating primary ovarian insufficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18-40
2. Menstrual cycle change more than 7 days at least 2 times,amenorrhea less than 6 months.
3. Sex hormone:bFSH>10u/L;or E2>80pg/ml.
4. AMH<1ng/ml.
5. Informed consent and truthfully answer the question.

Exclusion Criteria:

1. Dose not meet the inclusion criteria.
2. Genital tract malformation,congenital germinal aplasia, uterine amenorrhea and so on organic disease.
3. Endocrine diseases such Polycystic ovary syndrome、hyperprolactinemia 、dysfunctional uterine bleeding、low gonadotropin menstrual disorders and hyperthyreosis
4. Autoimmune disease patients:Hashimoto's thyroiditis,SLE,Primary chronic adrenal cortical insufficiency,Asthenic bulbar paralysis,Arthritis deformans,Idiopathic thrombocytopenic purpura, type I diabetes and so on.
5. Someone who have the following gynecological operation history: oophorocystectomy,ovarian drilling,wedgeshaped oophorectomy,adnexectomy,tubal resection,ligation of oviduct,pelvic abscess surgery,uterine arterial embolization.
6. Someone who have used reproductive toxicity drugs: tripterygium wilfordii,tripterygium hypoglaucum hutch,chemotherapeutics and so on.
7. A family history of ovarian failure.
8. Have receive hormone therapy in recent 3 months.
9. Pregnant or lactating women.
10. with serious heart,liver and kidney disease
11. With severe psychiatric disorders .
12. Have participated in other clinical trials in 3 months.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2016-04; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Anti-Mullerian hormone | 1year
  Anti-Mullerian hormone (AMH) is a gonadal hormone synthesized by granulose cells of the ovary and Sertoli cells of the testis. Anti-Mullerian hormone is used to facilitate the evaluation of intersex disorders and as a marker in ovarian reserve assessment in the infertility cases.

SECONDARY OUTCOMES:
Follicle stimulating hormone | 1year
  FSH is a gonadotropin, a glycoprotein polypeptide hormone. FSH is synthesized and secreted by the gonadotropic cells of the anterior pituitary gland,[1] and regulates the development, growth, pubertal maturation, and reproductive processes of the body.
Estrogen | 1year
  Estrogen is the primary female sex hormone as well as a medication.
Menopause rating scale | 1year
  The scale was designed and standardized as a self-administered scale to assess symptoms/complaints of aging women under different conditions, to evaluate the severity of symptoms over time, and to measure changes pre- and postmenopause replacement therapy
Menstrual Cycle | 1year
  The menstrual cycle is the regular natural change that occurs in the female reproductive system (specifically the uterus and ovaries) that makes pregnancy possible.

CONTACTS AND LOCATIONS:
Overall Officials: Hongyan Yang, professor, Study Chair — Guangzhou University of Traditional Chinese Medicine
Locations (1):
- Guangzhou University of Traditional Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided